CLINICAL TRIAL: NCT05037773
Title: Training Parents in an Elaborative Reminiscing Style to Boost Preschoolers' Development of Memory and Metacognition: A Randomized Controlled Study
Brief Title: Intervention Targeting Parental Reminiscing and Its Effects on Preschoolers' Memory and Metacognition
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Liege (Other)
Responsible Party: Principal Investigator, Christina Leonard, Principal Investigator, University of Liege
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: 1920-44
Record Dates: First submitted 2021-08-31; First posted 2021-09-08 (Actual); Last update posted 2021-09-08 (Actual); Status verified 2021-08

CONDITIONS: Child Development; Parent-Child Relations
Keywords: Typically developing preschoolers; Parental reminiscing; Memory; Metacognition

STUDY DESIGN:
Intervention Model Description: All participants receive the same intervention. However, Group 1 receives the intervention immediately after the baseline and Group 2 (i.e., the waiting-list group - acting as the control group -) receives the intervention after a second baseline assessment which is held after the completion of the Group 1 (i.e., approximatively 10 weeks later). Parent-child dyads were assigned to one of the 2 groups using a stratified randomization on children's age and when possible on children's gender.
  This design was chosen to check the specific efficiency of the intervention (i.e., which would result in no evolution for the Group 2 between the 2 baselines).
Who Masked: Outcomes Assessor
Masking Description: The outcome assessors (i.e., in charge of the baseline and post-intervention assessments) do not know to which group the participants belong.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): In this condition, the intervention is administered immediately after the baseline.
  Interventions: Behavioral: Intervention targeting parental reminiscing style
- Group 2 (waiting-list group) (Experimental): This group is both a control and an experimental group. Indeed, the intervention (i.e., the same as for group 1) is administered but after a second baseline which is held after the completion of the Group 1. This condition will allow to check the specific efficiency of the intervention.
  Interventions: Behavioral: Intervention targeting parental reminiscing style

INTERVENTIONS:
Behavioral: Intervention targeting parental reminiscing style — 8-session intervention (i.e., 1 session/week) targeting 3 main aspects of parental reminiscing: the promotion of child participation, the structure of discussions about the past and the content addressed during these discussions. Different learning techniques are used: psychoeducation, modeling and supervised practice.

SUMMARY:
This randomized controlled study aims to investigate the effects of an intervention targeting parental reminiscing style on preschoolers' memory (i.e., episodic and autobiographical) and metacognition (i.e., confidence judgment and memorability-based heuristic).

DETAILED DESCRIPTION:
It has been demonstrated that parental reminiscing plays an important role in preschoolers' cognitive development among which memory (Waters & al., 2019). Specifically, both correlational and interventional studies show that children of parents using a high-elaborative style during reminiscing (i.e., frequent, detailed and collaborative discussions about the past) recount their memories in a more detailed and coherent way (Wu & Jobson, 2019). Besides, some correlational studies (e.g., Langley et al., 2017) seem to also reveal an effect of parental reminiscing on children's ability to learn new information, as assessed in clinical neuropsychology by episodic memory tasks. However, the mechanisms underlying these influences are currently unclear. Indeed, several non-mutually exclusive hypotheses are frequently suggested (e.g., among which the development of metacognition (Rudek & Haden, 2005)) but, to date, have never been tested. Identifying these mechanisms could contribute to design interventions targeting parental reminiscing and to determine in which clinical contexts to use them. Currently, interventional studies in the field are scarce (for a review, see Corsano & Guidotti, 2019) and lack of consensus.

The primary aims of the present study are multiple. First, we aim to evaluate the effectiveness of a brief intervention program to improve the way parents reminisce with their child. After the intervention, we expect an increase in the frequency of use of the targeted behaviors and thus an increase in the level of parental elaboration. The second goal of this study is to explore the effects of the improvements in parental reminiscing style on children's memory skills, both autobiographical memory (i.e., ability to recount one's own memories) and episodic memory (i.e., ability to learn new information). Regarding autobiographical memory, we anticipate to replicate the results shown in other interventional studies (i.e., an increase in the amount of information reported by children at the end of the intervention; for a review, see Corsano & Guidotti, 2019). Regarding episodic memory, based on the results of correlational studies (e.g., Léonard et al., in prep), we anticipate after the intervention to show among children an improved ability to learn new information. Beyond these primary aims, secondary aims are also targeted in this study. Currently, the mechanisms underlying the relation between parental reminiscing and child's memory are still relatively unknown. A hypothesis that is frequently suggested is the development of metacognition (Rudek & Haden, 2005). One purpose of this study is to test this assumption by focusing on 2 metacognitive skills that develop during the preschool years: (a) the ability to make confidence judgments, (b) the ability to use the memorability-based heuristic. After the intervention, we expect children to make more accurate confidence judgments and to use more successfully the memorability-based heuristic to guide their memory decisions. Therefore, we may obtain information on the active ingredients of the relation between parental reminiscing and memory. Then, in an exploratory way, we explore whether such an intervention could improve parental cognitions as well as parents' perception of reminiscing with their child. We anticipate an improvement in parental cognitions and a more positive perception of reminiscing. Finally, we are interested in assessing parents' adherence to the intervention by exploring their feelings about its format, content and feasibility in daily life.

For all these purposes, a randomized controlled trial is currently being conducted. 2 experimental groups have been created and parent-child dyads were assigned to one of them using a stratified randomization on children's age and when possible on children's gender. Participants from both groups begin the study with an assessment of all variables of interest (i.e., baseline1). Immediately after this baseline assessment, participants from Group 1 receive the intervention. Participants from Group 2 (i.e., a waiting-list group acting as a control group) receive exactly the same intervention but later (i.e., after a second baseline assessment which is held after the completion of the intervention by the Group 1). Approximatively 2 weeks after the intervention, the dyads in each group undergo a post-intervention assessment (i.e., follow-up 1; similar to the baseline assessments). Besides, 6 months later, the Group 1 will participate in a follow-up session to check the persistence of the effects over time (i.e., follow-up 2). If the intervention is successful, this long-term follow-up may allow us to show either the maintenance of effects over time (e.g., an increase in parental elaboration) and/or the appearance of some effects (e.g., effects on child outcomes due to the time it takes for the improvement in parental style to have an effect on them).

In this study, all parents are provided with an 8-session intervention (i.e., 1 session/week) targeting different aspects of parental reminiscing: (a) the promotion of child participation (e.g., through parent's use of feedbacks), (b) the structure of reminiscing (e.g., parent's use of open-ended questions) and (c) the content addressed during reminiscing (e.g., contextual information). Parents learn to use the target behaviors through different standardized techniques: (a) psychoeducation, (b) modeling and (c) supervised practice. Due to Covid-19 epidemic, the intervention is held completely online (i.e., 4 e-learnings and 4 videoconferencing sessions).

ELIGIBILITY:
Inclusion Criteria:

* Children: French as mother tong
* Parent : be the parent who talks the most with the child (if both parents speak equally, the choice of the participating parent is left to them)

Exclusion Criteria:

* Children: major cognitive or language difficulties at the time of the study and attested by a neuropsychological or language assessment
* Children: actual medication that may lead to cognitive difficulties

Ages: 36 Months to 71 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2021-01-21 (Actual); Primary Completion 2022-01 (Estimated); Study Completion 2022-01 (Estimated)

PRIMARY OUTCOMES:
Parental reminiscing style | Group 1 : Baseline 1 (1 week before the intervention)
  Filmed parent-child discussion about a shared event of the previous day (as naturally as possible, without time constraint and in absence of the experimenter). These discussions will be transcribed for analysis with a specific coding scheme. Index : based on various raw scores, indexes will be computed.
Parental reminiscing style | Group 1 : Follow-up 1 (2 weeks after the intervention)
  Filmed parent-child discussion about a shared event of the previous day (as naturally as possible, without time constraint and in absence of the experimenter). These discussions will be transcribed for analysis with a specific coding scheme. Index : based on various raw scores, indexes will be computed.
Parental reminiscing style | Group 1 : Follow-up 2 (6 months after the intervention)
  Filmed parent-child discussion about a shared event of the previous day (as naturally as possible, without time constraint and in absence of the experimenter). These discussions will be transcribed for analysis with a specific coding scheme. Index : based on various raw scores, indexes will be computed.
Parental reminiscing style | Group 2 : Baseline 1 (10 weeks before the intervention)
  Filmed parent-child discussion about a shared event of the previous day (as naturally as possible, without time constraint and in absence of the experimenter). These discussions will be transcribed for analysis with a specific coding scheme. Index : based on various raw scores, indexes will be computed.
Parental reminiscing style | Group 2 : Baseline 2 (1 week before the intervention)
  Filmed parent-child discussion about a shared event of the previous day (as naturally as possible, without time constraint and in absence of the experimenter). These discussions will be transcribed for analysis with a specific coding scheme. Index : based on various raw scores, indexes will be computed.
Parental reminiscing style | Group 2 : Follow-up 1 (2 weeks after the intervention)
  Filmed parent-child discussion about a shared event of the previous day (as naturally as possible, without time constraint and in absence of the experimenter). These discussions will be transcribed for analysis with a specific coding scheme. Index : based on various raw scores, indexes will be computed.
Explicit knowledge about parental reminiscing | Group 1 : Baseline 1 (1 week before the intervention)
  10-item questionnaire aimed to assess parents' explicit knowledge about how to effectively discuss the past with their child (i.e., each item consists in a scenario and parents have to choose among different options which one would be the best way to interact with their child). 3 parallel versions of this questionnaire were created (i.e., order counterbalanced). Index : number of correct responses.
Explicit knowledge about parental reminiscing | Group 1 : Follow-up 1 (2 weeks after the intervention)
  10-item questionnaire aimed to assess parents' explicit knowledge about how to effectively discuss the past with their child (i.e., each item consists in a scenario and parents have to choose among different options which one would be the best way to interact with their child). 3 parallel versions of this questionnaire were created (i.e., order counterbalanced). Index : number of correct responses.
Explicit knowledge about parental reminiscing | Group 1 : Follow-up 2 (6 months after the intervention)
  10-item questionnaire aimed to assess parents' explicit knowledge about how to effectively discuss the past with their child (i.e., each item consists in a scenario and parents have to choose among different options which one would be the best way to interact with their child). 3 parallel versions of this questionnaire were created (i.e., order counterbalanced). Index : number of correct responses.
Explicit knowledge about parental reminiscing | Group 2 : Baseline 1 (10 weeks before the intervention)
  10-item questionnaire aimed to assess parents' explicit knowledge about how to effectively discuss the past with their child (i.e., each item consists in a scenario and parents have to choose among different options which one would be the best way to interact with their child). 3 parallel versions of this questionnaire were created (i.e., order counterbalanced). Index : number of correct responses.
Explicit knowledge about parental reminiscing | Group 2 : Baseline 2 (1 week before the intervention)
  10-item questionnaire aimed to assess parents' explicit knowledge about how to effectively discuss the past with their child (i.e., each item consists in a scenario and parents have to choose among different options which one would be the best way to interact with their child). 3 parallel versions of this questionnaire were created (i.e., order counterbalanced). Index : number of correct responses.
Explicit knowledge about parental reminiscing | Group 2 : Follow-up 1 (2 weeks after the intervention)
  10-item questionnaire aimed to assess parents' explicit knowledge about how to effectively discuss the past with their child (i.e., each item consists in a scenario and parents have to choose among different options which one would be the best way to interact with their child). 3 parallel versions of this questionnaire were created (i.e., order counterbalanced). Index : number of correct responses.
Children's autobiographical memory | Group 1 : Baseline 1 (1 week before the intervention)
  Retrieval of autobiographical memories cued by words (i.e., food, play, family, friend, happy, cry). 2 words/assessment (i.e., order counterbalanced). Children's production will be analyzed through a specific coding scheme. Index : the nature and the richness of information addressed by children.
Children's autobiographical memory | Group 1 : Follow-up 1 (2 weeks after the intervention)
  Retrieval of autobiographical memories cued by words (i.e., food, play, family, friend, happy, cry). 2 words/assessment (i.e., order counterbalanced). Children's production will be analyzed through a specific coding scheme. Index : the nature and the richness of information addressed by children.
Children's autobiographical memory | Group 1 : Follow-up 2 (6 months after the intervention)
  Retrieval of autobiographical memories cued by words (i.e., food, play, family, friend, happy, cry). 2 words/assessment (i.e., order counterbalanced). Children's production will be analyzed through a specific coding scheme. Index : the nature and the richness of information addressed by children.
Children's autobiographical memory | Group 2 : Baseline 1 (10 weeks before the intervention)
  Retrieval of autobiographical memories cued by words (i.e., food, play, family, friend, happy, cry). 2 words/assessment (i.e., order counterbalanced). Children's production will be analyzed through a specific coding scheme. Index : the nature and the richness of information addressed by children.
Children's autobiographical memory | Group 2 : Baseline 2 (1 week before the intervention)
  Retrieval of autobiographical memories cued by words (i.e., food, play, family, friend, happy, cry). 2 words/assessment (i.e., order counterbalanced). Children's production will be analyzed through a specific coding scheme. Index : the nature and the richness of information addressed by children.
Children's autobiographical memory | Group 2 : Follow-up 1 (2 weeks after the intervention)
  Retrieval of autobiographical memories cued by words (i.e., food, play, family, friend, happy, cry). 2 words/assessment (i.e., order counterbalanced). Children's production will be analyzed through a specific coding scheme. Index : the nature and the richness of information addressed by children.
Children's episodic memory (1) | Group 1 : Baseline 1 (1 week before the intervention)
  Assessment of children's ability to learn new information through the House Test (Picard et al., 2012) and 2 parallel versions created by our research team for this study (i.e., order counterbalanced). These tasks include an encoding phase and a retrieval phase in the form of free-recall and recognition after a 10-minute delay Index : number of correct responses at the free-recall task and the recognition task.
Children's episodic memory (1) | Group 1 : Follow-up 1 (2 weeks after the intervention)
  Assessment of children's ability to learn new information through the House Test (Picard et al., 2012) and 2 parallel versions created by our research team for this study (i.e., order counterbalanced). These tasks include an encoding phase and a retrieval phase in the form of free-recall and recognition after a 10-minute delay Index : number of correct responses at the free-recall task and the recognition task.
Children's episodic memory (1) | Group 1 : Follow-up 2 (6 months after the intervention)
  Assessment of children's ability to learn new information through the House Test (Picard et al., 2012) and 2 parallel versions created by our research team for this study (i.e., order counterbalanced). These tasks include an encoding phase and a retrieval phase in the form of free-recall and recognition after a 10-minute delay Index : number of correct responses at the free-recall task and the recognition task.
Children's episodic memory (1) | Group 2 : Baseline 1 (10 weeks before the intervention)
  Assessment of children's ability to learn new information through the House Test (Picard et al., 2012) and 2 parallel versions created by our research team for this study (i.e., order counterbalanced). These tasks include an encoding phase and a retrieval phase in the form of free-recall and recognition after a 10-minute delay Index : number of correct responses at the free-recall task and the recognition task.
Children's episodic memory (1) | Group 2 : Baseline 2 (1 week before the intervention)
  Assessment of children's ability to learn new information through the House Test (Picard et al., 2012) and 2 parallel versions created by our research team for this study (i.e., order counterbalanced). These tasks include an encoding phase and a retrieval phase in the form of free-recall and recognition after a 10-minute delay Index : number of correct responses at the free-recall task and the recognition task.
Children's episodic memory (1) | Group 2 : Follow-up 1 (2 weeks after the intervention)
  Assessment of children's ability to learn new information through the House Test (Picard et al., 2012) and 2 parallel versions created by our research team for this study (i.e., order counterbalanced). These tasks include an encoding phase and a retrieval phase in the form of free-recall and recognition after a 10-minute delay Index : number of correct responses at the free-recall task and the recognition task.
Children's episodic memory (2) | Group 1 : Baseline 1 (1 week before the intervention)
  Assessment of children's ability to learn new information through a story-recall task which consists of listening to a story (i.e., encoding phase) immediately followed by a true-false recognition. 3 comparable story-recall tasks were created (i.e., order counterbalanced). Index : a signal detection analysis (Macmillan & Creelman, 2005) will be performed to calculate sensitivity scores (i.e., reflecting children's ability to discriminate between studied information and lures).
Children's episodic memory (2) | Group 1 : Follow-up 1 (2 weeks after the intervention)
  Assessment of children's ability to learn new information through a story-recall task which consists of listening to a story (i.e., encoding phase) immediately followed by a true-false recognition. 3 comparable story-recall tasks were created (i.e., order counterbalanced). Index : a signal detection analysis (Macmillan & Creelman, 2005) will be performed to calculate sensitivity scores (i.e., reflecting children's ability to discriminate between studied information and lures).
Children's episodic memory (2) | Group 1 : Follow-up 2 (6 months after the intervention)
  Assessment of children's ability to learn new information through a story-recall task which consists of listening to a story (i.e., encoding phase) immediately followed by a true-false recognition. 3 comparable story-recall tasks were created (i.e., order counterbalanced). Index : a signal detection analysis (Macmillan & Creelman, 2005) will be performed to calculate sensitivity scores (i.e., reflecting children's ability to discriminate between studied information and lures).
Children's episodic memory (2) | Group 2 : Baseline 1 (10 weeks before the intervention)
  Assessment of children's ability to learn new information through a story-recall task which consists of listening to a story (i.e., encoding phase) immediately followed by a true-false recognition. 3 comparable story-recall tasks were created (i.e., order counterbalanced). Index : a signal detection analysis (Macmillan & Creelman, 2005) will be performed to calculate sensitivity scores (i.e., reflecting children's ability to discriminate between studied information and lures).
Children's episodic memory (2) | Group 2 : Baseline 2 (1 week before the intervention)
  Assessment of children's ability to learn new information through a story-recall task which consists of listening to a story (i.e., encoding phase) immediately followed by a true-false recognition. 3 comparable story-recall tasks were created (i.e., order counterbalanced). Index : a signal detection analysis (Macmillan & Creelman, 2005) will be performed to calculate sensitivity scores (i.e., reflecting children's ability to discriminate between studied information and lures).
Children's episodic memory (2) | Group 2 : Follow-up 1 (2 weeks after the intervention)
  Assessment of children's ability to learn new information through a story-recall task which consists of listening to a story (i.e., encoding phase) immediately followed by a true-false recognition. 3 comparable story-recall tasks were created (i.e., order counterbalanced). Index : a signal detection analysis (Macmillan & Creelman, 2005) will be performed to calculate sensitivity scores (i.e., reflecting children's ability to discriminate between studied information and lures).

SECONDARY OUTCOMES:
Children's confidence judgments | Group 1 : Baseline 1 (1 week before the intervention)
  Assessment of children's ability to make accurate confidence judgments when performing the aforementioned story-recall tasks. In these tasks, for each memory decision, children have to rate their confidence in their decisions through a 2-point pictorial scale (for a study using this method, see Geurten & Bastin, 2019). Index : the meta d'/d' ratio (Fleming & Lau, 2014) will be calculated to reflect children's ability to make accurate confidence judgments.
Children's confidence judgments | Group 1 : Follow-up 1 (2 weeks after the intervention)
  Assessment of children's ability to make accurate confidence judgments when performing the aforementioned story-recall tasks. In these tasks, for each memory decision, children have to rate their confidence in their decisions through a 2-point pictorial scale (for a study using this method, see Geurten & Bastin, 2019). Index : the meta d'/d' ratio (Fleming & Lau, 2014) will be calculated to reflect children's ability to make accurate confidence judgments.
Children's confidence judgments | Group 1 : Follow-up 2 (6 months after the intervention)
  Assessment of children's ability to make accurate confidence judgments when performing the aforementioned story-recall tasks. In these tasks, for each memory decision, children have to rate their confidence in their decisions through a 2-point pictorial scale (for a study using this method, see Geurten & Bastin, 2019). Index : the meta d'/d' ratio (Fleming & Lau, 2014) will be calculated to reflect children's ability to make accurate confidence judgments.
Children's confidence judgments | Group 2 : Baseline 1 (10 weeks before the intervention)
  Assessment of children's ability to make accurate confidence judgments when performing the aforementioned story-recall tasks. In these tasks, for each memory decision, children have to rate their confidence in their decisions through a 2-point pictorial scale (for a study using this method, see Geurten & Bastin, 2019). Index : the meta d'/d' ratio (Fleming & Lau, 2014) will be calculated to reflect children's ability to make accurate confidence judgments.
Children's confidence judgments | Group 2 : Baseline 2 (1 week before the intervention)
  Assessment of children's ability to make accurate confidence judgments when performing the aforementioned story-recall tasks. In these tasks, for each memory decision, children have to rate their confidence in their decisions through a 2-point pictorial scale (for a study using this method, see Geurten & Bastin, 2019). Index : the meta d'/d' ratio (Fleming & Lau, 2014) will be calculated to reflect children's ability to make accurate confidence judgments.
Children's confidence judgments | Group 2 : Follow-up 1 (2 weeks after the intervention)
  Assessment of children's ability to make accurate confidence judgments when performing the aforementioned story-recall tasks. In these tasks, for each memory decision, children have to rate their confidence in their decisions through a 2-point pictorial scale (for a study using this method, see Geurten & Bastin, 2019). Index : the meta d'/d' ratio (Fleming & Lau, 2014) will be calculated to reflect children's ability to make accurate confidence judgments.
Children's use of the memorability-based heuristic | Group 1 : Baseline 1 (1 week before the intervention)
  Assessment of children's use of the memorability-based heuristic when performing the aforementioned story-recall tasks. Indeed, this measure was allowed by the inclusion in each story of 8 low-memorable events and 8 high-memorable events. Children's use of the memorability-based heuristic was measured by contrasting their tendency to be more or less conservative in memory decisions for low-memorable versus high-memorable events. Index: a signal detection analysis (Macmillan & Creelman, 2005) will be performed to calculate response bias scores.
Children's use of the memorability-based heuristic | Group 1 : Follow-up 1 (2 weeks after the intervention)
  Assessment of children's use of the memorability-based heuristic when performing the aforementioned story-recall tasks. Indeed, this measure was allowed by the inclusion in each story of 8 low-memorable events and 8 high-memorable events. Children's use of the memorability-based heuristic was measured by contrasting their tendency to be more or less conservative in memory decisions for low-memorable versus high-memorable events. Index: a signal detection analysis (Macmillan & Creelman, 2005) will be performed to calculate response bias scores.
Children's use of the memorability-based heuristic | Group 1 : Follow-up 2 (6 months after the intervention)
  Assessment of children's use of the memorability-based heuristic when performing the aforementioned story-recall tasks. Indeed, this measure was allowed by the inclusion in each story of 8 low-memorable events and 8 high-memorable events. Children's use of the memorability-based heuristic was measured by contrasting their tendency to be more or less conservative in memory decisions for low-memorable versus high-memorable events. Index: a signal detection analysis (Macmillan & Creelman, 2005) will be performed to calculate response bias scores.
Children's use of the memorability-based heuristic | Group 2 : Baseline 1 (10 weeks before the intervention)
  Assessment of children's use of the memorability-based heuristic when performing the aforementioned story-recall tasks. Indeed, this measure was allowed by the inclusion in each story of 8 low-memorable events and 8 high-memorable events. Children's use of the memorability-based heuristic was measured by contrasting their tendency to be more or less conservative in memory decisions for low-memorable versus high-memorable events. Index: a signal detection analysis (Macmillan & Creelman, 2005) will be performed to calculate response bias scores.
Children's use of the memorability-based heuristic | Group 2 : Baseline 2 (1 week before the intervention)
  Assessment of children's use of the memorability-based heuristic when performing the aforementioned story-recall tasks. Indeed, this measure was allowed by the inclusion in each story of 8 low-memorable events and 8 high-memorable events. Children's use of the memorability-based heuristic was measured by contrasting their tendency to be more or less conservative in memory decisions for low-memorable versus high-memorable events. Index: a signal detection analysis (Macmillan & Creelman, 2005) will be performed to calculate response bias scores.
Children's use of the memorability-based heuristic | Group 2 : Follow-up 1 (2 weeks after the intervention)
  Assessment of children's use of the memorability-based heuristic when performing the aforementioned story-recall tasks. Indeed, this measure was allowed by the inclusion in each story of 8 low-memorable events and 8 high-memorable events. Children's use of the memorability-based heuristic was measured by contrasting their tendency to be more or less conservative in memory decisions for low-memorable versus high-memorable events. Index: a signal detection analysis (Macmillan & Creelman, 2005) will be performed to calculate response bias scores.

OTHER OUTCOMES:
Parents' perception of reminiscing with their child (exploratory) | Group 1 : Baseline 1 (1 week before intervention)
  The first 5 words that come to parents' mind when they think about the discussions they have with their child about school days. Index : the mean of valence of words (i.e., negative, neutral, positive) assessed by external judges.
Parents' perception of reminiscing with their child (exploratory) | Group 1 : Follow-up 1 (2 weeks after the intervention)
  The first 5 words that come to parents' mind when they think about the discussions they have with their child about school days. Index : the mean of valence of words (i.e., negative, neutral, positive) assessed by external judges.
Parents' perception of reminiscing with their child (exploratory) | Group 1 : Follow-up 2 (6 months after the intervention)
  The first 5 words that come to parents' mind when they think about the discussions they have with their child about school days. Index : the mean of valence of words (i.e., negative, neutral, positive) assessed by external judges.
Parents' perception of reminiscing with their child (exploratory) | Group 2 : Baseline 1 (10 weeks before the intervention)
  The first 5 words that come to parents' mind when they think about the discussions they have with their child about school days. Index : the mean of valence of words (i.e., negative, neutral, positive) assessed by external judges.
Parents' perception of reminiscing with their child (exploratory) | Group 2 : Baseline 2 (1 week before the intervention)
  The first 5 words that come to parents' mind when they think about the discussions they have with their child about school days. Index : the mean of valence of words (i.e., negative, neutral, positive) assessed by external judges.
Parents' perception of reminiscing with their child (exploratory) | Group 2 : Follow-up 1 (2 weeks after the intervention)
  The first 5 words that come to parents' mind when they think about the discussions they have with their child about school days. Index : the mean of valence of words (i.e., negative, neutral, positive) assessed by external judges.
Parenting cognitions (exploratory) | Group 1 : Baseline 1 (1 week before the intervention)
  Assessment of parenting cognitions as defined by Bornstein et al. (2018) through visual analogue scales (e.g., parental self-efficacy, parental satisfaction, parenting knowledge, ...). Index : position on visual analogue scales (from 0 to 10).
Parenting cognitions (exploratory) | Group 1 : Follow-up 1 (2 weeks after the intervention)
  Assessment of parenting cognitions as defined by Bornstein et al. (2018) through visual analogue scales (e.g., parental self-efficacy, parental satisfaction, parenting knowledge, ...). Index : position on visual analogue scales (from 0 to 10).
Parenting cognitions (exploratory) | Group 1 : Follow-up 2 (6 months after the intervention)
  Assessment of parenting cognitions as defined by Bornstein et al. (2018) through visual analogue scales (e.g., parental self-efficacy, parental satisfaction, parenting knowledge, ...). Index : position on visual analogue scales (from 0 to 10).
Parenting cognitions (exploratory) | Group 2 : Baseline 1 (10 weeks before the intervention)
  Assessment of parenting cognitions as defined by Bornstein et al. (2018) through visual analogue scales (e.g., parental self-efficacy, parental satisfaction, parenting knowledge, ...). Index : position on visual analogue scales (from 0 to 10).
Parenting cognitions (exploratory) | Group 2 : Baseline 2 (2 weeks before the intervention)
  Assessment of parenting cognitions as defined by Bornstein et al. (2018) through visual analogue scales (e.g., parental self-efficacy, parental satisfaction, parenting knowledge, ...). Index : position on visual analogue scales (from 0 to 10).
Parenting cognitions (exploratory) | Group 2 : Follow-up 1 (2 weeks after the intervention)
  Assessment of parenting cognitions as defined by Bornstein et al. (2018) through visual analogue scales (e.g., parental self-efficacy, parental satisfaction, parenting knowledge, ...). Index : position on visual analogue scales (from 0 to 10).
Parents' general feeling (exploratory) | Group 1 : Baseline 1 (1 week before the intervention)
  Visual analogue scales about parents' level of anxiety, depression, irritability and life satisfaction. Index : position on visual analogue scales (from 0 to 10).
Parents' general feeling (exploratory) | Group 1 : Follow-up 1 (2 weeks after the intervention)
  Visual analogue scales about parents' level of anxiety, depression, irritability and life satisfaction. Index : position on visual analogue scales (from 0 to 10).
Parents' general feeling (exploratory) | Group 1 : Follow-up 2 (6 months after the intervention)
  Visual analogue scales about parents' level of anxiety, depression, irritability and life satisfaction. Index : position on visual analogue scales (from 0 to 10).
Parents' general feeling (exploratory) | Group 2 : Baseline 1 (10 weeks before the intervention)
  Visual analogue scales about parents' level of anxiety, depression, irritability and life satisfaction. Index : position on visual analogue scales (from 0 to 10).
Parents' general feeling (exploratory) | Group 2 : Baseline 2 (1 week before the intervention)
  Visual analogue scales about parents' level of anxiety, depression, irritability and life satisfaction. Index : position on visual analogue scales (from 0 to 10).
Parents' general feeling (exploratory) | Group 2 : Follow-up 1 (2 weeks after the intervention)
  Visual analogue scales about parents' level of anxiety, depression, irritability and life satisfaction. Index : position on visual analogue scales (from 0 to 10).
Feasibility and adherence of the intervention (exploratory) | Group 1 : Follow-up 1 (2 weeks after the intervention)
  Online questionnaire in the form of visual analogue scales (e.g., measure of the degree of ease with which the parents apply the target behaviors in daily life) and open-ended questions (e.g., barriers to the daily use of the target behaviors). The drop-out rate will also be analyzed.
Feasibility and adherence of the intervention (exploratory) | Group 2 : Follow-up 1 (2 weeks after the intervention)
  Online questionnaire in the form of visual analogue scales (e.g., measure of the degree of ease with which the parents apply the target behaviors in daily life) and open-ended questions (e.g., barriers to the daily use of the target behaviors). The drop-out rate will also be analyzed.

CONTACTS AND LOCATIONS:
Overall Officials: Marie Geurten, Study Director — University of Liege; Sylvie Willems, Study Director — University of Liege
Locations (1):
- University of Liege, Liège, Belgium

IPD SHARING:
Plan to Share IPD: No
Data and analyses will be available from an online repository or from the principal investigator.

REFERENCES:
- [Background] Waters TEA, Camia C, Facompre CR, Fivush R. A meta-analytic examination of maternal reminiscing style: Elaboration, gender, and children's cognitive development. Psychol Bull. 2019 Nov;145(11):1082-1102. doi: 10.1037/bul0000211. PMID 31621348
- [Background] Wu Y, Jobson L. Maternal reminiscing and child autobiographical memory elaboration: A meta-analytic review. Dev Psychol. 2019 Dec;55(12):2505-2521. doi: 10.1037/dev0000821. Epub 2019 Sep 19. PMID 31535892
- [Background] Langley HA, Coffman JL, Ornstein PA. The Socialization of Children's Memory: Linking Maternal Conversational Style to the Development of Children's Autobiographical and Deliberate Memory Skills. J Cogn Dev. 2017;18(1):63-86. doi: 10.1080/15248372.2015.1135800. Epub 2016 Sep 10. PMID 29270083
- [Background] Rudek DJ, Haden CA. Mothers' and Preschoolers' Mental State Language During Reminiscing Over Time. Merrill Palmer Q. 2005;51(4):557-583. doi: 10.1353/mpq.2005.0026
- [Background] Corsano P, Guidotti L. Parents' reminiscing training in typically developing and 'at-risk' children: a review. Early Child Dev Care. 2019; 189(1): 143-156. doin: 10.1080/03004430.2017.1289518
- [Background] Geurten M, Bastin C. Behaviors speak louder than explicit reports: Implicit metacognition in 2.5-year-old children. Dev Sci. 2019 Mar;22(2):e12742. doi: 10.1111/desc.12742. Epub 2018 Sep 19. PMID 30159971
- [Background] Bornstein MH, Putnick DL, Suwalsky JTD. Parenting cognitions --> parenting practices --> child adjustment? The standard model. Dev Psychopathol. 2018 May;30(2):399-416. doi: 10.1017/S0954579417000931. Epub 2017 Jun 19. PMID 28625208
- [Derived] Leonard C, Geurten M, Willems S. Parental reminiscing training and preschoolers' memory and metacognition: A randomized controlled trial. Dev Psychol. 2023 Jul;59(7):1167-1180. doi: 10.1037/dev0001514. Epub 2023 May 18. PMID 37199921